CLINICAL TRIAL: NCT06024317
Title: Leveraging Community Health Workers and a Responsive Digital Health System to Improve Rates and Timeliness of Child Well Visits in the First Year of Life
Brief Title: Leveraging Community Health Workers and a Digital Health System to Improve the Timeliness of Child Well Visits
Acronym: MINT-II/HKW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Duke University (Other); Emory University (Other); University of North Carolina (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Jan Ostermann, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00120675
Record Dates: First submitted 2023-08-28; First posted 2023-09-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Short Message Service (SMS); Incentives; Knowledge, Attitudes, Practice; Preventive Services
Keywords: Timeliness; Digital Health; Community Health Workers; Tanzania; Low and middle-income country; SMS reminder; Conditional incentive; Preventive services; Children
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: This type 1 effectiveness-implementation hybrid study uses a cluster-randomized trial design to evaluate intervention effectiveness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Huduma Kwa Wakati) (Experimental): Within the catchment areas of 40 health facilities, 40 communities ("clusters"; 1 per catchment area) will be assigned to the intervention arm. 40 communities ("clusters"; 1 per catchment area) will be assigned to the control arm. 10 pregnant women in their last trimester of pregnancy will be enrolled from each cluster. Women enrolled from intervention clusters will receive all components of the Huduma Kwa Wakati intervention.
  Interventions: Behavioral: Huduma Kwa Wakati - Knowledge Intervention; Behavioral: Huduma Kwa Wakati - Reminders; Behavioral: Huduma Kwa Wakati - Incentives; Behavioral: Huduma Kwa Wakati - Service notifications
- Control (Standard of care) (No Intervention): Within the catchment areas of 40 health facilities, 40 communities ("clusters"; 1 per catchment area) will be assigned to the intervention arm. 40 communities ("clusters"; 1 per catchment area) will be assigned to the control arm. 10 pregnant women in their last trimester of pregnancy will be enrolled from each cluster. Women enrolled from control arm will receive baseline and follow-up assessments only.

INTERVENTIONS:
Behavioral: Huduma Kwa Wakati - Knowledge Intervention — Counseling scripts assessing and addressing child health-related knowledge gaps
  Arms: Intervention arm (Huduma Kwa Wakati)
Behavioral: Huduma Kwa Wakati - Reminders — Reminders of upcoming well visit due dates, sent to the mother's mobile phone
  Arms: Intervention arm (Huduma Kwa Wakati)
Behavioral: Huduma Kwa Wakati - Incentives — Conditional incentives for timely service receipt, tailored to each child's well visit schedule
  Arms: Intervention arm (Huduma Kwa Wakati)
Behavioral: Huduma Kwa Wakati - Service notifications — Service notifications (e.g., related to stockouts or service non-availability), sent to the mother's mobile phone
  Arms: Intervention arm (Huduma Kwa Wakati)

SUMMARY:
The goal of this cluster-randomized type 1 effectiveness implementation hybrid trial is to evaluate whether a community health worker led, integrated digital health intervention (Huduma Kwa Wakati; "Timely Services" in Kiswahili) can improve rates of timely well visits and receipt of key recommended preventive interventions among children in their first year of life. The hypothesis is that Huduma Kwa Wakati will improve the timeliness and rates of completion of child well visits and receipt of recommended preventive services before age 1 year, compared to the standard of care. Researchers will compare outcomes among children enrolled from intervention clusters and no-intervention comparison clusters. Outcomes will also be compared to a cross-sectional retrospective comparison sample. This study will address the lack of rigorous evidence on the effectiveness of a community-based digital health intervention for promoting rates and timeliness of preventive service receipt among children from sub-Saharan Africa, and identify implementation strategies to facilitate the deployment of integrated community-based digital health interventions in low- and middle-income country settings.

DETAILED DESCRIPTION:
Background and Objective:

In Tanzania, only 68% of children receive key recommended preventive health interventions within their first year of life. Prior research identified substantial rural-urban disparities in rates and timeliness of preventive service receipt in Tanzania, with children in rural settings being more like to receive delayed or no services. This type 1 effectiveness implementation hybrid study will evaluate the effect of Huduma Kwa Wakati ("Timely Services" in Kiswahili), a community-based, integrated digital health intervention, on the timeliness of child well visits and receipt of recommended preventive services in children's first year of life. The intervention combines a knowledge intervention, mobile phone-based reminders, and incentives with the goal to promote timely service receipt.

Methods:

The study will be conducted in the catchment areas of 40 rural health facilities in two predominantly rural regions in Tanzania. From each catchment area, three cohorts of mother-child dyads, one retrospective cohort and two prospective cohorts, will be enrolled into the study. The prospective cohort, comprising mothers from eighty communities ("clusters") within these catchment areas, will be randomized to an intervention or control arm. The timeliness (primary outcome) and coverage (secondary outcome) of child well visits will be observed for 1200 children (800 prospective children and 400 retrospective children). Details of the clinical trial refer to the prospective cohort of 800 mother-child dyads. Study logs, fidelity checklists, quantitative surveys, child health records, and qualitative interviews with mothers and key informants will be used to inform the five constructs of the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework. Results will be used to develop an implementation blueprint that can guide future adaptations, sustainability, and scale-up of Huduma Kwa Wakati.

Hypothesis:

The hypothesis is that Huduma Kwa Wakati is effective for increasing the timeliness of child well visits and rates of preventive services receipt before age 1 year compared to the standard of care.

Expected impact:

This study will address the lack of rigorous evidence on the effectiveness of a community-based digital health intervention for promoting rates and timeliness of recommended health service receipt among children from sub-Saharan Africa, and identify implementation strategies to facilitate the deployment of integrated interventions in low- and middle-income country settings.

ELIGIBILITY:
Inclusion Criteria for the Cross-sectional sample:

* mothers of children ages 12-23 months
* residing in the sampling area

Inclusion Criteria for the Longitudinal sample:

* pregnant women in their last trimester of pregnancy
* residing in the sampling area
* expected to reside in the sampling area until the child reaches age 1 year

Exclusion Criteria:

* Women who are not living in catchment areas of participating health facilities (which routinely provide maternal and child health services). Facilities must be operational, must have at least 2 community health workers, and must have reported at least 100 pregnancies or births in the year prior to study implementation.)

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Delay in days (continuous) for the child well visit due at age 14 weeks | Assessed during the endline survey, an average follow-up period of 1 year
  The average number of days between the due date of the 14 week well visit and the date on which the child actually attends this visit. Dates abstracted from the child's health book.

SECONDARY OUTCOMES:
Delay > 28 days (binary) for the child well visit due at age 14 weeks | Assessed during the endline survey, an average follow-up period of 1 year
  The percentage of participants with a delay >28 days between the visit due date (at age 14 weeks) and the date on which the visit was attended. Dates abstracted from the child's health book.

OTHER OUTCOMES:
Receipt of all recommended services during the child's first year of life (binary) | Assessed during the endline survey, an average follow-up period of 1 year
  The percentage of children who attended all visits and received all services recommended by age 1 year. Coverage abstracted from the child's health book.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ostermann, PhD, Principal Investigator — University of South Carolina
Locations (1):
- National Institute for Medical Research, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No
The data from this study will be available from the National Institute for Medical Research, Muhimbili Research Centre, Tanzania, but restrictions apply that are governed by consent forms and data transfer agreements. Data may be made available by the authors upon reasonable request and with permission of the National Medical Research Review Committee at the National Institute for Medical Research (NIMR) in Tanzania.

REFERENCES:
- [Background] Yelverton V, Hair NL, Ghosh SH, Mfinanga SG, Ngadaya E, Baumgartner JN, Ostermann J, Vasudevan L. Beyond coverage: Rural-urban disparities in the timeliness of childhood vaccinations in Tanzania. Vaccine. 2022 Sep 2;40(37):5483-5493. doi: 10.1016/j.vaccine.2022.07.020. Epub 2022 Aug 10. PMID 35961796
- [Background] Vasudevan L, Baumgartner JN, Moses S, Ngadaya E, Mfinanga SG, Ostermann J. Parental concerns and uptake of childhood vaccines in rural Tanzania - a mixed methods study. BMC Public Health. 2020 Oct 20;20(1):1573. doi: 10.1186/s12889-020-09598-1. PMID 33081744
- [Background] Ostermann J, Vasudevan L, Baumgartner JN, Ngadaya E, Mfinanga SG. Do mobile phone-based reminders and conditional financial transfers improve the timeliness of childhood vaccinations in Tanzania? Study protocol for a quasi-randomized controlled trial. Trials. 2019 Jul 4;20(1):397. doi: 10.1186/s13063-019-3430-4. PMID 31272487
- [Background] Ostermann J, Hair NL, Moses S, Ngadaya E, Godfrey Mfinanga S, Brown DS, Noel Baumgartner J, Vasudevan L. Is the intention to vaccinate enough? Systematic variation in the value of timely vaccinations and preferences for monetary vs non-monetary incentives among pregnant women in southern Tanzania. Vaccine X. 2023 Jan 23;13:100266. doi: 10.1016/j.jvacx.2023.100266. eCollection 2023 Apr. PMID 36814594
- [Background] Vasudevan L, Ostermann J, Moses SM, Ngadaya E, Mfinanga SG. Patterns of Mobile Phone Ownership and Use Among Pregnant Women in Southern Tanzania: Cross-Sectional Survey. JMIR Mhealth Uhealth. 2020 Apr 8;8(4):e17122. doi: 10.2196/17122. PMID 32267240
- [Derived] Vasudevan L, Ostermann J, Thielman N, Baumgartner JN, Solomon D, Mosses A, Hobbie A, Hair NL, Liang C, van Zwetselaar M, Mfinanga S, Ngadaya E. Leveraging Community Health Workers and a Responsive Digital Health System to Improve Vaccination Coverage and Timeliness in Resource-Limited Settings: Protocol for a Cluster Randomized Type 1 Effectiveness-Implementation Hybrid Study. JMIR Res Protoc. 2024 Jan 12;13:e52523. doi: 10.2196/52523. PMID 38214956